CLINICAL TRIAL: NCT05673525
Title: A Clinical Trial of the Transcatheter Aortic Valve Implantation System With a Prospective, Multi-Center, One-Arm Approach to Evaluate the Efficacy and Safety in the Treatment of Patients With Severe Aortic Stenosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Chief, Department of Structural Heart DiseaseAffiliation, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOKA-2022-03
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Aortic Stenosis
Keywords: Heart Valve Disease; Cardiovascular Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Cardiovascular Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Device: Transcatheter Aortic Valve Implantation (KOKA-VALVE)

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (KOKA-VALVE) — Transcatheter Aortic Valve Implantation

SUMMARY:
A Clinical Trial of the Transcatheter Aortic Valve Implantation System with a Prospective, Multi-Center, One-Arm Approach to Evaluate the Efficacy and Safety in the Treatment of Patients with Severe Aortic Stenosis

DETAILED DESCRIPTION:
This trial consists of two parts. Part I, the Feasibility trial: 10-12 patients with severe aortic stenosis who meet inclusion/exclusion criteria and are at high surgical risk or not suitable for conventional surgical valve replacement are selected at no more than 5 centers for implantation of an aortic valve by transcatheter aortic valve replacement (KOKA-VALVE) to achieve treatment of aortic valve disease in subjects. All-cause mortality at 30 days after implantation is used as the primary endpoint, and the immediate postoperative device success and surgical success, major cardiovascular adverse events at 1 year after implantation, transvalvular pressure difference at 30 days and 12 months after implantation, degree of orifice regurgitation, degree of perivalvular leakage, improvement in NYHA cardiac function, and improvement in quality of survival are used as the secondary endpoints to supplementarily evaluate the safety and feasibility of this product. It also provides experience and reference for further Part II confirmatory trials and applications to ensure safe conduct of confirmatory trials. Subjects in the feasibility trial may continue to be followed up at 6 months after implantation and 12 months after implantation after completion of the one-month postoperative follow-up. All subjects will also continue to be followed up by telephone at 24, 36, 48, and 60 months after implantation.

Part II, the Confirmatory Trial: Designed with a prospective, multi-center, one-arm approach. 131 patients with severe aortic stenosis who meet inclusion/non-exclusion criteria and are at high surgical risk or unsuitable for conventional surgical valve replacement are implanted with an aortic valve by transcatheter aortic valve replacement (KOKA-VALVE) to achieve treatment of aortic valve disease in subjects. All-cause mortality at 30 days after implantation is used as the primary endpoint, and the immediate postoperative device success and surgical success, major cardiovascular adverse events at 1 year after implantation, transvalvular pressure difference at 30 days and 12 months after implantation, degree of orifice regurgitation, degree of perivalvular leakage, improvement in NYHA cardiac function, and improvement in quality of survival are used as the secondary endpoints to supplementarily evaluate the safety and feasibility of this product.

All patients will be followed up before discharge, 30 days, 6 months, and 12 months after implantation after product implantation. All subjects will be followed up by telephone at 24 months, 36 months, 48 months and 60 months after implantation.

The study will be conducted at multiple clinical trial sites nationwide, and 131 subjects will be enrolled in the confirmatory trial. The enrollment and treatment status of the subjects will be recorded during the study, and the subjects will be followed up before discharge, 6 months after implantation, and 12 months after implantation, and the data will be compiled for registration and declaration.

All subjects will be followed up by telephone at 24 months, 36 months, 48 months, and 60 months after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Contraindication to surgery, or high risk for surgery (STS ≥ 8%) as assessed by the heart team; or other circumstances that make surgical valve replacement inappropriate.
* Age ≥65 years.
* Patients with symptomatic severe aortic stenosis (mean aortic transvalvular gradient by echocardiography ≥40 mmHg (1 mmHg=0.133 kPa), or transaortic flow velocity ≥4.0 m/s, or aortic valve orifice area <0.8 cm2, or effective aortic orifice area index <0.5 cm2 /m2).
* The subjects have been informed of the nature of this study, understand the purpose of the clinical trial, and voluntarily participate in and sign the informed consent form.

Exclusion Criteria:

* Life expectancy less than 1 year after implantation of the prosthetic valve.
* Patients had an acute heart attack within 1 month, or had a coronary stent or a pacing device implantation within 1 month, or had any therapeutic cardiac surgery within 1 month.
* Patients with aortic root anatomy and lesion that are not suitable for prosthetic valve implantation.
* Combined with severe insufficiency or stenosis of other valves and requiring surgical treatment.
* Hematologic cachexia, including leukopenia (WBC <3×10^9 /L), acute anemia (HB <90 g/L), thrombocytopenia (PLT <50 × 10^9 /L), bleeding constitution, and coagulation disorders.
* Untreated coronary artery disease requiring hematologic reconstruction.
* Hypertrophic obstructive cardiomyopathy.
* Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) <20%.
* Severe right ventricular insufficiency.
* The existent of intracardiac masses, thrombi or superfluous organisms by echocardiography.
* Patients who cannot tolerate anticoagulation or antiplatelet therapy.
* Patients had cerebrovascular event (CVA), including ischemic stroke and hemorrhagic stroke within 3 months.
* Decompensation of renal insufficiency.
* Active infective endocarditis or other active infection.
* Untreated conduction system disease requiring pacemaker implantation.
* Currently participating in an investigational drug or another device study that has not completed its primary endpoints or would clinically interfere with the endpoint of this study.
* Other circumstances that are assessed by the investigator to be unsuitable for interventional aortic valve therapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months postoperatively
  Cumulative all-cause mortality at 12 months postoperatively

SECONDARY OUTCOMES:
Transvalvular Gradient | 30 days and 12 months postoperatively
  Transvalvular Gradients at 30 days and 12 months postoperatively
Aortic Regurgitation Degree | 30 days and 12 months postoperatively
  Aortic Regurgitation Degree at 30 days and 12 months postoperatively
Perivalvular Leakage | 30 days and 12 months postoperatively
  Perivalvular Leakage at 30 days and 12 months postoperatively
Cardiac Function | 30 days and 12 months postoperatively
  The rate of New York Heart Association (NYHA) Function Class at 30 days and 12 months postoperatively
Quality of Survival | 30 days and 12 months postoperatively
  The score of EQ-5D at 30 days and 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Structral Heart Disease Center, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No